CLINICAL TRIAL: NCT05424809
Title: Feasibility and Preliminary Effectiveness of a Shared Decision-making Process in a Tertiary University Hospital: Protocol of a Pilot Randomized Clinical Trial
Brief Title: Feasibility and Preliminary Effectiveness of a Shared Decision-making Process
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Karla Salas Gama, Dr Karla Salas-Gama - Quality Department, Hospital Vall d'Hebron, Hospital Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PR(AG)148/2022
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Clinical Decision Making; Patient-Centered Care; Obesity; Chronic Kidney Diseases
MeSH Terms: conditions — Obesity; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared decision-making model (Experimental): In the intervention group, the shared decision-making model will be carried out. This model was proposed and designed through a participatory and deliberative process.
  Interventions: Behavioral: Shared decision-making model
- Usual care (No Intervention): Information without an estructured shared decision-making model

INTERVENTIONS:
Behavioral: Shared decision-making model — The model is based on a person-centred care process, where an exchange of information is carried out between the health professional and the patient to make the best decision that is consistent with the person's values and preferences.
  A six-stage process constitutes the model: 1) Identificacion of the decision point, 2) design of a specific patient decision aid, 3) identification of possible barriers and ways to overcome them, 4) training for professionals, 5) 3-steps implementation of shared decision-making in clinical practice, 6) evaluation
  Arms: Shared decision-making model

SUMMARY:
Background: Shared decision-making is a process where health professionals and patients work together through conversation and using tools to make the best possible decision for the person. Patient decision aids provide information based on the best available evidence, support the deliberative process, and further help clarifies individual patient values and preferences. Incorporating shared decision-making in clinical practice is challenging.

Hypothesis: A proposed shared decision-making implementation model is feasible and improves patients' knowledge of possible treatment options, as well as patients' perception and degree of satisfaction with the decision-making process.

Objective: To evaluate the feasibility and preliminary effectiveness of implementing a shared decision-making model in a tertiary university hospital.

Methods: It is proposed to carry out a pilot randomized clinical study (ratio 1:1), with two arms, in parallel, open, single center. Adult patients from two clinical processes will be included: a) Obesity (treatment options: bariatric surgery or medical management (healthy habits +/- pharmacological treatment), and b) Advanced Chronic Kidney Disease (ACKD) (treatment options: hemodialysis, peritoneal dialysis, or conservative treatment).

Since it is a pilot study, the investigators estimated a random sample of between 20 to 40 participants per intervention group and control group (total sample 40 to 80 per pathology) would be needed. The intervention group will carry out the shared decision-making model, and the control group will receive the usual clinical practice with detailed information from a health professional.

The primary outcomes of interest to be evaluated are a) feasibility; b) quality of the decision and the decision-making process.

DETAILED DESCRIPTION:
Background: Shared decision-making is a process where health professionals and patients work together through conversation and using tools to make the best possible decision for the person. Patient decision aids provide information based on the best available evidence, support the deliberative process, and further help clarifies individual patient values and preferences. Incorporating shared decision-making in clinical practice is challenging. Some studies have analyzed the implementation of shared decision-making in specific clinical processes. However, the investigators have only been able to identify one study, still in progress, that plans to implement and evaluate the integration of a shared decision-making program in a university hospital.

Hypothesis: The proposed shared decision-making implementation model is feasible and improves patients' knowledge of possible treatment options, as well as patients' perception and degree of satisfaction with the decision-making process.

Objective: To evaluate the feasibility and preliminary effectiveness of implementing a shared decision-making model in a tertiary university hospital.

Methods: It is proposed to carry out a pilot randomized clinical study (ratio 1:1), with two arms, in parallel, open, single center. The guidelines of the 2010 CONSORT statement for reporting randomized trials will be followed. Adult patients from two clinical processes will be included: a) Obesity (treatment options: bariatric surgery or medical management (healthy habits +/- pharmacological treatment), and b) Advanced Chronic Kidney Disease (ACKD) (treatment options to decide: hemodialysis, peritoneal dialysis, or conservative treatment).

Since it is a pilot study, the investigators estimated a random sample of between 20 to 40 participants per intervention group and control group (total sample 40 to 80 per pathology) would be needed. The intervention group will carry out the shared decision-making model, and the control group will receive the usual clinical practice with detailed information from a health professional.

The outcomes of interest to be evaluated are a) feasibility (defined by the number of patients in the intervention group who agree to participate in a shared decision-making process and who complete the entire study process); b) quality of the decision and the decision-making process (defined by the degree of knowledge, scale of satisfaction with the decision, quality of the process, decisional conflict and perception of information and inclusion in the process).

The recruitment of patients will begin in May 2022. The assignment of patients in Obesity will be carried out from the Agenda Service, where a person outside the research team will randomly assign each patient to the first visit of the intervention group or control group. In ACKD, the assignment will be randomly through the REDCap computer program. The coded collection of variables will also be carried out through the REDCap program.

ELIGIBILITY:
Inclusion Criteria Obesity:

* Adult patients, between 18 and 60 years old, Spanish or Catalan speakers, who have scheduled a visit to the obesity clinic.
* BMI≥40Kg/m2 or ≥35kg/m2 with major associated comorbidities, likely to improve after weight loss
* Presence of morbid obesity established for at least five years
* Absence of endocrine disorders that cause obesity
* Favorable psychiatric-psychological evaluation
* Informed consent to participate in the study after having received all the necessary information (oral and written)

Exclusion Criteria Obesity:

* Patient with cognitive impairment that does not allow for a shared decision-making process.
* Unstable organic disease limiting the probability of success and benefit of participation in the obesity unit program.
* Patients previously operated on bariatric surgery
* Clinical contraindications included in the general criteria of the Bariatric Surgery Protocol of the Hospital Universitari Vall d'Hebron
* Clinical contraindications for pharmacological treatment according to technical date of GLP-1 analogues (Trulicity, Ozempic, Victoza, Saxenda)

Inclusion Criteria ACKD:

* Adult patients aged 18 or over who speak Spanish or Catalan who have a scheduled visit to the ACKD clinic.
* Advanced chronic kidney disease (GFR ≤20ml/min) that requires assessment of the start of renal replacement therapy through any dialysis, transplant or conservative treatment.
* Informed consent to participate in the study after having received all the necessary information (oral and written)

Exclusion Criteria ACKD:

* Having previously performed any modality of renal replacement therapy.
* Patient with cognitive impairment that does not allow for a shared decision-making process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-11-23 (Estimated); Study Completion 2022-12-23 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the decision-making model | 4-6 weeks
  The number of patients in the intervention group agreed to participate in a shared decision-making process and complete the entire process until answering the questionnaires. A value of ≥80% of the intervention group will be considered viable
Preliminary effectiveness - Knowledge | 4-6 weeks
  Measured through multiple-choice questions proposed by the study researchers. We will measure the number of correct answers in both groups
Preliminary effectiveness - Satisfaction with decision | 4-6 weeks
  Measured with the self-reported Satisfaction With Decision scale (SWDs) (6 items with 5-item Likert scales)
Preliminary effectiveness - Perception of shared decision-making process | 4-6 weeks
  Measures patients' perceptions of how clinicians' performance fits the shared decision-making process. We will use the self-reported 9-item Shared Decision-Making Questionnaire (9 items with 6-item Likert scale)
Preliminary effectiveness - Decisional conflict | 4-6 weeks
  Measured with the self-reported Decisional Conflict Scale (16 items with 5-item Likert scale)
Preliminary effectiveness - Perception of participation in the decision-making process | 4-6 weeks
  Measured with the CollaboRATE scale (3 item self-report questions, range from 0 to 7

SECONDARY OUTCOMES:
Decision made | 4-6 weeks
  Number of participants that choose one option:
  * Obesity group: surgical intervention vs medical treatment
  * ACKD group: hemodialysis vs peritoneal dialysis vs conservative care
Duration of each medical visit | 4-6 weeks
  We will measure, in minutes, the total time of clinical encounters for both groups
Number of visits necessary until the final decision is made | 4-6 weeks
  number of visits

CONTACTS AND LOCATIONS:
Overall Officials: Karla Salas Gama, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fearns N, Kelly J, Callaghan M, Graham K, Loudon K, Harbour R, Santesso N, McFarlane E, Thornton J, Treweek S. What do patients and the public know about clinical practice guidelines and what do they want from them? A qualitative study. BMC Health Serv Res. 2016 Feb 24;16:74. doi: 10.1186/s12913-016-1319-4. PMID 27121606
- [Background] Stacey D, Legare F, Lewis K, Barry MJ, Bennett CL, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2017 Apr 12;4(4):CD001431. doi: 10.1002/14651858.CD001431.pub5. PMID 28402085
- [Background] Elwyn G, Frosch D, Thomson R, Joseph-Williams N, Lloyd A, Kinnersley P, Cording E, Tomson D, Dodd C, Rollnick S, Edwards A, Barry M. Shared decision making: a model for clinical practice. J Gen Intern Med. 2012 Oct;27(10):1361-7. doi: 10.1007/s11606-012-2077-6. Epub 2012 May 23. PMID 22618581
- [Background] Legare F, Adekpedjou R, Stacey D, Turcotte S, Kryworuchko J, Graham ID, Lyddiatt A, Politi MC, Thomson R, Elwyn G, Donner-Banzhoff N. Interventions for increasing the use of shared decision making by healthcare professionals. Cochrane Database Syst Rev. 2018 Jul 19;7(7):CD006732. doi: 10.1002/14651858.CD006732.pub4. PMID 30025154
- [Background] Sondergaard SR, Madsen PH, Hilberg O, Jensen KM, Olling K, Steffensen KD. A prospective cohort study of shared decision making in lung cancer diagnostics: Impact of using a patient decision aid. Patient Educ Couns. 2019 Nov;102(11):1961-1968. doi: 10.1016/j.pec.2019.05.018. Epub 2019 May 16. PMID 31129012
- [Background] Steffensen KD, Vinter M, Cruger D, Dankl K, Coulter A, Stuart B, Berry LL. Lessons in Integrating Shared Decision-Making Into Cancer Care. J Oncol Pract. 2018 Apr;14(4):229-235. doi: 10.1200/JOP.18.00019. PMID 29641952
- [Background] Danner M, Geiger F, Wehkamp K, Rueffer JU, Kuch C, Sundmacher L, Skjelbakken T, Rummer A, Novelli A, Debrouwere M, Scheibler F; SHARE TO CARE (S2C) Project Team. Making shared decision-making (SDM) a reality: protocol of a large-scale long-term SDM implementation programme at a Northern German University Hospital. BMJ Open. 2020 Oct 10;10(10):e037575. doi: 10.1136/bmjopen-2020-037575. PMID 33039998
- [Background] Chabrera C, Areal J, Font A, Caro M, Bonet M, Zabalegui A. [Spanish version of the Satisfaction With Decision scale: cross-cultural adaptation, validity and reliability]. Enferm Clin. 2015 May-Jun;25(3):117-23. doi: 10.1016/j.enfcli.2015.02.005. Epub 2015 Apr 25. Spanish. PMID 25921323
- [Background] De las Cuevas C, Perestelo-Perez L, Rivero-Santana A, Cebolla-Marti A, Scholl I, Harter M. Validation of the Spanish version of the 9-item Shared Decision-Making Questionnaire. Health Expect. 2015 Dec;18(6):2143-53. doi: 10.1111/hex.12183. Epub 2014 Mar 5. PMID 24593044
- [Background] Urrutia M, Campos S, O'Connor A. [Validation of a Spanish version of the Decisional Conflict scale]. Rev Med Chil. 2008 Nov;136(11):1439-47. doi: 10.4067/s0034-98872008001100010. Spanish. PMID 19301775
- [Background] Bravo P, Contreras A, Dois A, Villarroel L. [Adapting and validating the generic instrument CollaboRATE to measure women's participation in health related decision-making during the reproductive process]. Aten Primaria. 2018 May;50(5):274-281. doi: 10.1016/j.aprim.2017.04.003. Epub 2017 Jul 29. Spanish. PMID 28760344